CLINICAL TRIAL: NCT05994027
Title: Attachment & Child Health (ATTACH™) Online Platform: Helping Children Vulnerable to Early Adversity
Brief Title: ATTACH™ Online Platform: Helping Children Vulnerable to Early Adversity
Acronym: ATTACH™
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Nicole Letourneau, Chair in Parent-Infant Mental Health. Professor, Faculty of Nursing & Cumming School of Medicine (Pediatrics, Psychiatry & Community Health Sciences), Director of RESOLVE Alberta, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB20-0903-Online
Record Dates: First submitted 2023-07-22; First posted 2023-08-16 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Parent-Child Relations
Keywords: Parent Child Interaction Quality; Parental Reflective Function; Child Development; Online platform

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATTACH™ Online Platform Parenting Program (Other): A quasi-experimental design was selected to more closely approximate service delivery models in agencies that do not typically employ control groups.
  Given promising findings (from seven ATTACH™ pilot studies), a randomized controlled trial design, even employing wait-list controls, was deemed unacceptable and even unethical by patients, healthcare professionals, and health system administrators in engagement activities surrounding the preparation of this proposal.
  Interventions: Behavioral: ATTACH™ Online Platform Parenting Program

INTERVENTIONS:
Behavioral: ATTACH™ Online Platform Parenting Program — ATTACH Online Platform: Preserving and promoting optimal RF in parents who are experiencing adversities, enables parents to appropriately attribute affective states to their children and respond accurately to meet their children's needs, thus promoting sensitive/ responsive parent-child relationships.

SUMMARY:
Addressing the impact of early childhood adversity (e.g., family violence, parental depression, and low income) can promote children's mental health and development, giving children the best start in life and reducing societal health inequities. Family violence, depression, and low income undermine parent-child relationship quality linked to mental health and developmental problems in children that tend to persist over the lifespan. Parents' reflective function (RF), i.e., the capacity to understand their own and their child's thoughts, feelings, and mental states, can strengthen parent-child relationships and buffer the negative impacts of early adversity on children. Investigators have developed and tested an effective intervention program called ATTACH™ (Attachment and Child Health) for parents and their preschool-aged children at-risk of early adversity. In research with 90 families, investigators found the intervention significantly improved RF, parent-child relationship quality, and children's mental health and development. When COVID-19 prevented in-person intervention at the same time as demand soared for ATTACH™, investigators developed and pilot tested (n=10) an Online platform or "platform" with our community partners, including parents, to deliver the program virtually. The purpose of the study is to propose an effective implementation hybrid (EIH) Type II study of the ATTACH™ Online platform. Co-primary objectives evaluate clinical intervention effectiveness and implementation strategy feasibility of the ATTACH™ Online platform in naturalistic, real-world settings delivered by community partner agencies serving families affected by early adversity in Alberta.

DETAILED DESCRIPTION:
Methods: This effectiveness-implementation hybrid (EIH) Type II study is an innovative clinical trial comprised of a quasi-experimental design evaluation of the community-agency delivered ATTACH™ Online platform (with measurement pre-intervention, immediately post-intervention, and three months postintervention) as well as an examination of implementation feasibility via Normalization Process Theory. Investigators will work with 100 parents and children (aged newborn to 36 months).

Objective 1: Employing innovative clinical trial quasi-experimental methods, the effectiveness of the ATTACH™ Online platform will be evaluated on: (1a) children's mental health and development (primary outcome), parent-child relationship quality, and parental reflective function (secondary outcomes) immediately and three months after the intervention, (1b) different patient populations (for whom the program works best/worst), and (1c) health professionals' adherence to the clinical intervention protocol via fidelity assessment. For these objectives, investigators will intervene with 100 new families, a sufficiently powered n to detect minimum d=.5 (from pilot data and accounting for attrition) for pre-intervention/post-intervention differences in children's mental health and development.

Objective 2: Using qualitative methods, the feasibility of implementation of the ATTACH™ Online platform will be evaluated via (2a) knowledge of users' (patients/parents, health care professionals, and administrators) perceptions and experiences of the ATTACH™ Online platform, (2b) ATTACH™ Online platform uptake, and (2c) ATTACH™ Online platform implementation benefits, facilitators, barriers, and challenges. For these objectives, investigators will interview knowledge users (patients/parents, health care professionals, and administrators (n≈60)) until data saturation using Normalization Process Theory.

Study Setting： include 10 Alberta agencies (technically 9, as one agency operates two shelters) serving culturally diverse clients (i.e., Caucasian as well as Black, Indigenous, People of Colour; BIPOC) and immigrants affected by family violence, depression, and low-income. The agencies including Brenda Strafford Centre, Catholic Social Services, Children, Families, and Community Services, Central Alberta Women's Emergency Shelter, Discovery House (Women's Shelter), Highbanks, Home Next Door*, Hull Social Services, Julietta's Place, La Salle Second Stage Shelter, Catholic Social Services and WINGS of Providence.

ELIGIBILITY:
Inclusion Criteria:

* parents with children between birth to 32 months of age (our age ceiling is 36 months, based on selection of age-platformropriate tools for assessing children's health and development );
* parents who agree to participate in the ATTACH™ Online platform program consisting of 10 weeks of additional, concurrent, one-hour per week parent training sessions;
* parents who agree to bring a co-parent for 2 of the 10 sessions (when possible).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Children's Mental Health and Development | Change from baseline ASQ-3 scores immediately after completion of intervention and at 3 months.
  The Ages and Stages Questionnaire 3rd Edition (ASQ - 3) is a series of parent-completed questionnaires to assess child development in 5 domains namely communication, gross motor, fine motor, problem-solving, and personal-social skills. There are 21 versions for different age groups 21 ranging from 1 to 66 months, with 6 questions in each domain asking if the child can or cannot do age-appropriate tasks. Adding up items in each domain provides a total score for that domain. Summing up the total scores for each domain yields the total score (out of 60). Scores range from 0-60 and higher scores are indicative of healthier outcomes.

SECONDARY OUTCOMES:
Parent-Child Relationship Quality | Change from baseline PCITS scores immediately after completion of intervention and at 3 months.
  The Parent Child Interaction Teaching Scale (PCITS) is an observational binary measure of interactions in parent-child teaching situations to measure parent-child interaction quality in infants 36 months or younger. Considered as the gold standard, PCITS consists of 73 items categorized into 6 subscales including parental sensitivity to cues, responsiveness to distress, growth fostering, and cognitive growth fostering, and infant clarity of cues and responsiveness to parent. Certified coders code the items either as yes or no; Yes responses are then summed to yield a total score for each sub-scale. Final PCITS scores include total scores for each subscale, parent total, child total, and parent-child total scores, along with total parent contingency and child contingency scores. The observation of teaching interaction typically takes 5 minutes. Scale range from 0 - 73. A higher score means a better outcome, i.e. higher quality of parent-child interaction.
Parental Reflective Function (RF) | Change from baseline PRFQ scores immediately after completion of intervention and at 3 months.
  The Parental Reflective Function Questionnaire (PRFQ) is an 18-item measure of parental RF, with subscales assessing: (a) Pre-mentalizing subscale, (b) Certainty in Mental States subscale, and (c) Interest and Curiosity subscale. Scores from each sub-scale range from 1 to 7. Higher scores indicate higher levels of parental RF. The PRFQ has good internal consistency (.7-.84) and takes 5 minutes to complete. Pilot testing revealed the PRFQ detected intervention impacts and was acceptable to patients. In our other work, investigators show that scores on the PRFQ associate significantly (p<.05) with the gold standard Parental Development Interview coded with Fonagy's 11-point scale. Given the gold standard requires 1-2 hours per patient interview, followed by 1 hour to check automated transcriptions, and 3 hours of coding per interview (~6 hours total), the use of the PRFQ reduces patient burden, costs and is feasible to implement in agencies.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Letourneau, PhD RN, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anis L, Letourneau N, Benzies K, Ewashen C, Hart MJ. Effect of the Attachment and Child Health Parent Training Program on Parent-Child Interaction Quality and Child Development. Can J Nurs Res. 2020 Jun;52(2):157-168. doi: 10.1177/0844562119899004. Epub 2020 Jan 30. PMID 32000509
- [Result] Ross KM, Cole S, Sanghera H, Anis L, Hart M, Letourneau N. The ATTACH program and immune cell gene expression profiles in mothers and children: A pilot randomized controlled trial. Brain Behav Immun Health. 2021 Oct 2;18:100358. doi: 10.1016/j.bbih.2021.100358. eCollection 2021 Dec. PMID 34647106
- [Result] Letourneau N, Anis L, Novick J, Pohl C, Ntanda H, Hart M. Impacts of the Attachment and Child Health (ATTACHTM) Parenting Program on Mothers and Their Children at Risk of Maltreatment: Phase 2 Results. Int J Environ Res Public Health. 2023 Feb 9;20(4):3078. doi: 10.3390/ijerph20043078. PMID 36833770
- [Result] Anis L, Letourneau N, Ross KM, Hart M, Graham I, Lalonde S, Varro S, Baldwin A, Soulsby A, Majnemer A, Donnelly C, Piotrowski C, Collier C, Lindeman C, Goldowitz D, Isaac D, Thomson D, Serre D, Citro E, Zimmermann G, Pliszka H, Mann J, Baumann J, Piekarski J, Dalton JA, Johnson-Green J, Wood K, Bruce M, Santana M, Mayer M, Gould M, Kobor M, Flowers M, Haywood M, Koerner M, Parker N, Muhajarine N, Fairie P, Chrishti R, Perry R, Merrill S, Pociuk S, StephanieTaylor, Cole S, Murphy T, Marchment T, Xavier V, Shajani Z, West Z. Study protocol for Attachment & Child Health (ATTACHTM) program: promoting vulnerable Children's health at scale. BMC Pediatr. 2022 Aug 19;22(1):491. doi: 10.1186/s12887-022-03439-3. PMID 35986306
- [Result] Letourneau N, Anis L, Ntanda H, Novick J, Steele M, Steele H, Hart M. Attachment & Child Health (ATTACH) pilot trials: Effect of parental reflective function intervention for families affected by toxic stress. Infant Ment Health J. 2020 Jul;41(4):445-462. doi: 10.1002/imhj.21833. Epub 2020 Jun 13. PMID 32533796
- [Result] Anis L, Ross K, Ntanda H, Hart M, Letourneau N. Effect of Attachment and Child Health (ATTACHTM) Parenting Program on Parent-Infant Attachment, Parental Reflective Function, and Parental Depression. Int J Environ Res Public Health. 2022 Jul 10;19(14):8425. doi: 10.3390/ijerph19148425. PMID 35886276
- [Result] Squires J, Bricker D, Potter L. Revision of a parent-completed development screening tool: Ages and Stages Questionnaires. J Pediatr Psychol. 1997 Jun;22(3):313-28. doi: 10.1093/jpepsy/22.3.313. PMID 9212550
- [Result] Luyten P, Mayes LC, Nijssens L, Fonagy P. The parental reflective functioning questionnaire: Development and preliminary validation. PLoS One. 2017 May 4;12(5):e0176218. doi: 10.1371/journal.pone.0176218. eCollection 2017. PMID 28472162
- [Result] Letourneau NL, Tryphonopoulos PD, Novick J, Hart JM, Giesbrecht G, Oxford ML. Nursing Child Assessment Satellite Training Parent-Child Interaction Scales: Comparing American and Canadian Normative and High-Risk Samples. J Pediatr Nurs. 2018 May-Jun;40:47-57. doi: 10.1016/j.pedn.2018.02.016. Epub 2018 Mar 22. PMID 29776479
- [Result] Anis L, Benzies KM, Ewashen C, Hart MJ, Letourneau N. Fidelity Assessment Checklist Development for Community Nursing Research in Early Childhood. Front Public Health. 2021 May 14;9:582950. doi: 10.3389/fpubh.2021.582950. eCollection 2021. PMID 34055705
- [Derived] Letourneau N, Anis L, Cui C, Graham ID, Ross K, Nixon K, Reimer J, Pilipchuk M, Wang E, Lalonde S, Varro S, Santana MJ, Stewart-Tufescu A, Soulsby A, Tiedemann B, Hill L, Beks T, Hart M. Study protocol for assessing the effectiveness, implementation fidelity and uptake of attachment & child health (ATTACH) Online: helping children vulnerable to early adversity. BMC Pediatr. 2025 Apr 9;25(1):280. doi: 10.1186/s12887-024-05232-w. PMID 40205561